CLINICAL TRIAL: NCT07116655
Title: Improving Mental Health Treatment Engagement of Patients With Comorbid Chronic Diseases: A Randomized Controlled Evaluation of the Feasibility and Preliminary Effectiveness of a Single-Session Solution-Focused Consultation (SSC) in a Community Setting
Brief Title: Feasibility Study of Single-session Solution Focused Consultation to Enhance Treatment Engagement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanyang Technological University (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB-2024-777
Record Dates: First submitted 2025-08-06; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-03

CONDITIONS: Treatment Engagement
Keywords: treatment engagement; chronic physical health problems; comorbid mental health problems; single-session intervention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Control Group (Active Comparator): Single-session supportive therapy based approach
  Interventions: Behavioral: Single-session supportive intervention
- Intervention Group (Experimental): Single-session solution-focused therapy based approach
  Interventions: Behavioral: Single-session solution focused consultation

INTERVENTIONS:
Behavioral: Single-session solution focused consultation — In the SSC, the interventionist first sets expectations, explaining that the session is a means of providing short-term support. The interventionist will then praise the participant for agreeing to receive support and introduce the Action Plan, which will guide the session's structure. The interventionist will then work with the participant to (1) identify a specific, modifiable issue they are facing; (2) use the "miracle question" to envision their ideal outcome where the problem is resolved, and rates their current proximity to that; (3) determine the "smallest possible step" they can take towards this outcome through a scaling exercise; and (4) develop a personalized action plan that leverage on their current resources to begin addressing the problem. Upon ending the SSC, the interventionist writes a personalized note to the participant, highlighting their strengths and expressing confidence in their ability to follow through.
  Arms: Intervention Group
Behavioral: Single-session supportive intervention — In the supportive consultation session, the interventionist will allow the participant to decide what they wish to discuss during the session and listen empathetically, validate their feelings and offer reassurance to the patient. The exact wording or questions will vary depending on the client's needs and sharing.
  Arms: Active Control Group

SUMMARY:
This research aims to explore whether a single-session solution-focused consultation (SSC) can increase mental health service engagement among patients with comorbid chronic physical diseases and mental health problems (CPDMHP).

ELIGIBILITY:
Inclusion Criteria: 1. A history of one or more chronic physical diseases based on the Ministry of Health (Singapore) Chronic Disease Management Programme guidelines; 2. A score of 5 or more on the Patient Health Questionnaire (PHQ-9) or Generalized Anxiety Disorder-7 (GAD-7); 3. Not currently engaged in formal mental health service; 4. Conversant in the English language; 5. Receiving treatment in a community healthcare setting

Exclusion Criteria: 1. A history of psychosis, intellectual disability, or pervasive developmental disorders

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Treatment Engagement - Uptake | Post-intervention (immediate)
  Endorsement of interest in referral for mental health services or follow-up session with interventionist
Treatment engagement - Attendance | 2-weeks post-intervention
  Attendance at intake session for mental health services or follow-up session with interventionist
Feasibility - Intervention Completion Rate | Post-intervention (immediate)
  Completion of intervention action plans
Acceptability - Usefulness of intervention | Post-intervention (immediate)
  Single item measure on helpfulness of consultation in addressing concern/s
Acceptability - Satisfaction with outcome | Post-intervention (immediate)
  Single item measure on how satisfied they are with the intervention's outcome

SECONDARY OUTCOMES:
Perceived agency | From baseline to post-intervention (immediate)
  State Hope Scale (SHS) - Pathways Subscale
Hope | From baseline to post-intervention (immediate) and two-week post intervention
  Beck's Hopelessness Scale (BHS-4)

OTHER OUTCOMES:
Depression | From baseline to two-weeks post intervention
  Patient's Health Questionnaire (PHQ-9)
Anxiety | From baseline to two-weeks post intervention
  Generalized Anxiety Disorder (GAD-7)
Change readiness | From baseline to post-intervention (immediate) and two-week post intervention
  Readiness Ruler
Life satisfaction | From baseline to two-week post intervention
  Single-item measuring satisfaction with life
Perceived current health status | From baseline to two-week post intervention
  Single-item measuring perceived current health status

CONTACTS AND LOCATIONS:
Locations (1):
- Renal Health Services, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided